CLINICAL TRIAL: NCT02897739
Title: Pathogenesis of Acute Stress Induced (Tako-tsubo) Cardiomyopathy: Energy Shut-Down or Intense Inflammation? The TERRIFIC Study
Brief Title: Pathogenesis of Acute Stress Induced (Tako-tsubo) Cardiomyopathy: Energy Shut-Down or Intense Inflammation?
Acronym: TERRIFIC
Status: Completed | Type: Observational
Sponsor: University of Aberdeen (Other)
Collaborators: NHS Grampian (Other Government)
Responsible Party: Sponsor
Other Study IDs: 14/NS/1068
Record Dates: First submitted 2016-03-24; First posted 2016-09-13 (Estimated); Last update posted 2019-05-08 (Actual); Status verified 2019-05

CONDITIONS: Tako-tsubo Cardiomyopathy
MeSH Terms: conditions — Takotsubo Cardiomyopathy | interventions — Magnetic Resonance Spectroscopy

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 4 Months
Biospecimen Retention: Samples With DNA — EDTA blood samples, EDTA Plasma and Serum to be retained.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- TTC Patients: Patients diagnosed with Tako-tsubo cardiomyopathy.
  Interventions: Procedure: Magnetic resonance imaging; Biological: Acute Inflammatory Activation study; Radiation: PET CT; Behavioral: Psychological assessment
- Health Volunteers: Participants who have normal hearts.
  Interventions: Procedure: Magnetic resonance imaging; Biological: Acute Inflammatory Activation study; Radiation: PET CT; Behavioral: Psychological assessment

INTERVENTIONS:
Procedure: Magnetic resonance imaging — Cardiac MRI and short MRI following USPIO infusion
Biological: Acute Inflammatory Activation study — Blood sampling for exploration of type and level of inflammatory response
Radiation: PET CT — PET study for metabolic pathway study
Behavioral: Psychological assessment — Assessment by a psychologist

SUMMARY:
Tako Tsubo Cardiomyopathy (TTC), also known as "Broken Heart Syndrome", is a disorder of the heart that occurs most commonly in women (although it occasionally occurs in men) and is usually related to a stressful event. Symptoms are often similar to a heart attack, and include chest pain and shortness of breath. Although Tako Tsubo Cardiomyopathy is not a new medical condition, it has not been widely recognised until the last decade. Currently the investigators don't have an exact understanding of how or why the heart is affected in this way, and so the investigators are conducting a study to help understand what causes Tako Tsubo Cardiomyopathy.

DETAILED DESCRIPTION:
The investigators aim to study the reciprocal modulation of fatty acids and glucose metabolism in the Tako Tsubo Cardiomyopathy physiology, in both humans and an animal model, and to investigate which metabolic pathway is preferentially adopted by acute Tako Tsubo Cardiomyopathy myocytes during this severe functional shut down with largely preserved variability. The human model will be used to determine the preferential stimulated uptake of glucose/fatty acids under optimal metabolic conditions for each (hyperinsulineamic euglycemic clamp for 18F-Fludeoxyglucose (18F-FDG) and fasting for 14Fluorine-18Fluoro-6-Thia-Heptadecanoic Acid (18F-FTHA cardiac Positron Emission Tomography)). In the rat model the investigators will examine both the metabolic tracer uptake (using micro Positron Emission Tomography-Computed Tomography) as well as the downstream modulation of the two metabolic pathways (transcriptional regulators, mitochondrial respiration, expression of the uncoupling proteins, levels of Adenosine Triphosphate generation and reactive oxygen species production).

The investigators aim to test the hypothesis that inflammation plays a pivotal role in the pathophysiology of this condition by further exploring: 1) In the rat model define time course, extent and subtypes of cellular infiltrate, 2) In the rat model of Tako Tsubo Cardiomyopathy, demonstrate the presence of inflammatory macrophages using in-vivo Ultrasmall Superparamagnetic Iron Oxide-cardiac magnetic resonance imaging and whether this relates to numbers and types of macrophages present as determined by immunohistochemical analysis, 3) In clinical patients, define the time course of specific peripheral blood monocyte subsets and the serum levels of inflammatory cytokines versus matched controls and 4) In clinical patients, establish the compartmentalisation of tissue macrophages in the left ventricle its time course resolution using Ultrasmall Superparamagnetic Iron Oxide-enhanced cardiac magnetic resonance.

The investigators will assess the psycho-emotional factors involved in Tako Tsubo Cardiomyopathy given that in the majority of cases intense emotional trauma is immediately preceding onset.

ELIGIBILITY:
Inclusion Criteria:

* All patients diagnosed with TTC in the past 12 days, able to give consent and who have not lost capacity of consent between the time of diagnosis (usually made at coronary catheterisation, for which they are consented clinically) and time of being approached for inclusion in the study.
* Age and gender matched healthy controls willing to participate and able to give consent.

Exclusion Criteria:

* Unwillingness to participate
* Patients with contraindications to MR scanning
* Pregnant or breast-feeding women

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients who have been diagnosed with Tako-tsubo Cardiomyopathy Healthy volunteers
Sampling Method: Non-Probability Sample
Enrollment: 77 (Actual)
Dates: Start 2015-08 (Actual); Primary Completion 2019-03 (Actual); Study Completion 2019-03 (Actual)

PRIMARY OUTCOMES:
Cardiac Inflammation as measured by Cardiac Magnetic Resonance Imaging | Three years
  As measured by cardiac MRI

SECONDARY OUTCOMES:
Evidence of psycho-emotional factors following intense physical or emotional stress as measured by Hospital Anxiety and Depression Scale | Three years
  As measured by psychiatric interview
Evidence of alterations of the metabolism of myocardium by Cardiac Positron Emission Tomography | Three years
  As measured by PET CT
Systemic Inflammation as measured by inflammatory markers | Three years
  As measured by inflammatory markers

CONTACTS AND LOCATIONS:
Overall Officials: Dana Dawson, MD, MRCP, Principal Investigator — University of Aberdeen
Locations (1):
- Cardiac Research Office, Aberdeen, Aberdeenshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Prasad A, Lerman A, Rihal CS. Apical ballooning syndrome (Tako-Tsubo or stress cardiomyopathy): a mimic of acute myocardial infarction. Am Heart J. 2008 Mar;155(3):408-17. doi: 10.1016/j.ahj.2007.11.008. Epub 2008 Jan 31. PMID 18294473
- [Background] Gianni M, Dentali F, Grandi AM, Sumner G, Hiralal R, Lonn E. Apical ballooning syndrome or takotsubo cardiomyopathy: a systematic review. Eur Heart J. 2006 Jul;27(13):1523-9. doi: 10.1093/eurheartj/ehl032. Epub 2006 May 23. PMID 16720686
- [Background] Neil C, Nguyen TH, Kucia A, Crouch B, Sverdlov A, Chirkov Y, Mahadavan G, Selvanayagam J, Dawson D, Beltrame J, Zeitz C, Unger S, Redpath T, Frenneaux M, Horowitz J. Slowly resolving global myocardial inflammation/oedema in Tako-Tsubo cardiomyopathy: evidence from T2-weighted cardiac MRI. Heart. 2012 Sep;98(17):1278-84. doi: 10.1136/heartjnl-2011-301481. Epub 2012 Jul 11. PMID 22791656
- [Background] Sharkey SW, Windenburg DC, Lesser JR, Maron MS, Hauser RG, Lesser JN, Haas TS, Hodges JS, Maron BJ. Natural history and expansive clinical profile of stress (tako-tsubo) cardiomyopathy. J Am Coll Cardiol. 2010 Jan 26;55(4):333-41. doi: 10.1016/j.jacc.2009.08.057. PMID 20117439
- [Background] Abraham J, Mudd JO, Kapur NK, Klein K, Champion HC, Wittstein IS. Stress cardiomyopathy after intravenous administration of catecholamines and beta-receptor agonists. J Am Coll Cardiol. 2009 Apr 14;53(15):1320-5. doi: 10.1016/j.jacc.2009.02.020. PMID 19358948
- [Background] Nef HM, Mollmann H, Akashi YJ, Hamm CW. Mechanisms of stress (Takotsubo) cardiomyopathy. Nat Rev Cardiol. 2010 Apr;7(4):187-93. doi: 10.1038/nrcardio.2010.16. Epub 2010 Mar 2. PMID 20195267
- [Background] Elesber AA, Prasad A, Lennon RJ, Wright RS, Lerman A, Rihal CS. Four-year recurrence rate and prognosis of the apical ballooning syndrome. J Am Coll Cardiol. 2007 Jul 31;50(5):448-52. doi: 10.1016/j.jacc.2007.03.050. Epub 2007 Jul 16. PMID 17662398
- [Background] Neubauer S, Horn M, Naumann A, Tian R, Hu K, Laser M, Friedrich J, Gaudron P, Schnackerz K, Ingwall JS, et al. Impairment of energy metabolism in intact residual myocardium of rat hearts with chronic myocardial infarction. J Clin Invest. 1995 Mar;95(3):1092-100. doi: 10.1172/JCI117756. PMID 7883957
- [Background] Dawson DK, Neil CJ, Henning A, Cameron D, Jagpal B, Bruce M, Horowitz J, Frenneaux MP. The Authors Reply. JACC Cardiovasc Imaging. 2016 May;9(5):633. doi: 10.1016/j.jcmg.2015.02.032. Epub 2016 Feb 17. No abstract available. PMID 26897679
- [Background] Feola M, Chauvie S, Rosso GL, Biggi A, Ribichini F, Bobbio M. Reversible impairment of coronary flow reserve in takotsubo cardiomyopathy: a myocardial PET study. J Nucl Cardiol. 2008 Nov-Dec;15(6):811-7. doi: 10.1007/BF03007363. Epub 2008 Jul 31. PMID 18984457
- [Background] Yoshida T, Hibino T, Kako N, Murai S, Oguri M, Kato K, Yajima K, Ohte N, Yokoi K, Kimura G. A pathophysiologic study of tako-tsubo cardiomyopathy with F-18 fluorodeoxyglucose positron emission tomography. Eur Heart J. 2007 Nov;28(21):2598-604. doi: 10.1093/eurheartj/ehm401. Epub 2007 Oct 7. PMID 17921529
- [Background] Ibrahim T, Nekolla SG, Langwieser N, Rischpler C, Groha P, Laugwitz KL, Schwaiger M. Simultaneous positron emission tomography/magnetic resonance imaging identifies sustained regional abnormalities in cardiac metabolism and function in stress-induced transient midventricular ballooning syndrome: a variant of Takotsubo cardiomyopathy. Circulation. 2012 Nov 20;126(21):e324-6. doi: 10.1161/CIRCULATIONAHA.112.134346. No abstract available. PMID 23169256
- [Background] Gerber BL, Ordoubadi FF, Wijns W, Vanoverschelde JL, Knuuti MJ, Janier M, Melon P, Blanksma PK, Bol A, Bax JJ, Melin JA, Camici PG. Positron emission tomography using(18)F-fluoro-deoxyglucose and euglycaemic hyperinsulinaemic glucose clamp: optimal criteria for the prediction of recovery of post-ischaemic left ventricular dysfunction. Results from the European Community Concerted Action Multicenter study on use of(18)F-fluoro-deoxyglucose Positron Emission Tomography for the Detection of Myocardial Viability. Eur Heart J. 2001 Sep;22(18):1691-701. doi: 10.1053/euhj.2000.2585. PMID 11511119
- [Background] Herrero P, Peterson LR, McGill JB, Matthew S, Lesniak D, Dence C, Gropler RJ. Increased myocardial fatty acid metabolism in patients with type 1 diabetes mellitus. J Am Coll Cardiol. 2006 Feb 7;47(3):598-604. doi: 10.1016/j.jacc.2005.09.030. Epub 2006 Jan 18. PMID 16458143
- [Background] Kurisu S, Inoue I, Kawagoe T, Ishihara M, Shimatani Y, Nishioka K, Umemura T, Nakamura S, Yoshida M, Sato H. Myocardial perfusion and fatty acid metabolism in patients with tako-tsubo-like left ventricular dysfunction. J Am Coll Cardiol. 2003 Mar 5;41(5):743-8. doi: 10.1016/s0735-1097(02)02924-8. PMID 12628716
- [Background] Wittstein IS, Thiemann DR, Lima JA, Baughman KL, Schulman SP, Gerstenblith G, Wu KC, Rade JJ, Bivalacqua TJ, Champion HC. Neurohumoral features of myocardial stunning due to sudden emotional stress. N Engl J Med. 2005 Feb 10;352(6):539-48. doi: 10.1056/NEJMoa043046. PMID 15703419
- [Background] Paur H, Wright PT, Sikkel MB, Tranter MH, Mansfield C, O'Gara P, Stuckey DJ, Nikolaev VO, Diakonov I, Pannell L, Gong H, Sun H, Peters NS, Petrou M, Zheng Z, Gorelik J, Lyon AR, Harding SE. High levels of circulating epinephrine trigger apical cardiodepression in a beta2-adrenergic receptor/Gi-dependent manner: a new model of Takotsubo cardiomyopathy. Circulation. 2012 Aug 7;126(6):697-706. doi: 10.1161/CIRCULATIONAHA.112.111591. Epub 2012 Jun 25. PMID 22732314
- [Background] Shao Y, Redfors B, Scharin Tang M, Mollmann H, Troidl C, Szardien S, Hamm C, Nef H, Boren J, Omerovic E. Novel rat model reveals important roles of beta-adrenoreceptors in stress-induced cardiomyopathy. Int J Cardiol. 2013 Oct 3;168(3):1943-50. doi: 10.1016/j.ijcard.2012.12.092. Epub 2013 Jan 26. PMID 23357048
- [Background] Nef HM, Mollmann H, Kostin S, Troidl C, Voss S, Weber M, Dill T, Rolf A, Brandt R, Hamm CW, Elsasser A. Tako-Tsubo cardiomyopathy: intraindividual structural analysis in the acute phase and after functional recovery. Eur Heart J. 2007 Oct;28(20):2456-64. doi: 10.1093/eurheartj/ehl570. Epub 2007 Mar 29. PMID 17395683
- [Background] Ziegler-Heitbrock L, Ancuta P, Crowe S, Dalod M, Grau V, Hart DN, Leenen PJ, Liu YJ, MacPherson G, Randolph GJ, Scherberich J, Schmitz J, Shortman K, Sozzani S, Strobl H, Zembala M, Austyn JM, Lutz MB. Nomenclature of monocytes and dendritic cells in blood. Blood. 2010 Oct 21;116(16):e74-80. doi: 10.1182/blood-2010-02-258558. Epub 2010 Jul 13. PMID 20628149
- [Background] Gill JM, Saligan L, Woods S, Page G. PTSD is associated with an excess of inflammatory immune activities. Perspect Psychiatr Care. 2009 Oct;45(4):262-77. doi: 10.1111/j.1744-6163.2009.00229.x. PMID 19780999
- [Background] Alam SR, Shah AS, Richards J, Lang NN, Barnes G, Joshi N, MacGillivray T, McKillop G, Mirsadraee S, Payne J, Fox KA, Henriksen P, Newby DE, Semple SI. Ultrasmall superparamagnetic particles of iron oxide in patients with acute myocardial infarction: early clinical experience. Circ Cardiovasc Imaging. 2012 Sep 1;5(5):559-65. doi: 10.1161/CIRCIMAGING.112.974907. Epub 2012 Aug 8. PMID 22875883
- [Background] Yilmaz A, Dengler MA, van der Kuip H, Yildiz H, Rosch S, Klumpp S, Klingel K, Kandolf R, Helluy X, Hiller KH, Jakob PM, Sechtem U. Imaging of myocardial infarction using ultrasmall superparamagnetic iron oxide nanoparticles: a human study using a multi-parametric cardiovascular magnetic resonance imaging approach. Eur Heart J. 2013 Feb;34(6):462-75. doi: 10.1093/eurheartj/ehs366. Epub 2012 Oct 26. PMID 23103659
- [Background] Paternostro G, Camici PG, Lammerstma AA, Marinho N, Baliga RR, Kooner JS, Radda GK, Ferrannini E. Cardiac and skeletal muscle insulin resistance in patients with coronary heart disease. A study with positron emission tomography. J Clin Invest. 1996 Nov 1;98(9):2094-9. doi: 10.1172/JCI119015. PMID 8903329
- [Background] Chen X, Lee G, Maher BS, Fanous AH, Chen J, Zhao Z, Guo A, van den Oord E, Sullivan PF, Shi J, Levinson DF, Gejman PV, Sanders A, Duan J, Owen MJ, Craddock NJ, O'Donovan MC, Blackman J, Lewis D, Kirov GK, Qin W, Schwab S, Wildenauer D, Chowdari K, Nimgaonkar V, Straub RE, Weinberger DR, O'Neill FA, Walsh D, Bronstein M, Darvasi A, Lencz T, Malhotra AK, Rujescu D, Giegling I, Werge T, Hansen T, Ingason A, Noethen MM, Rietschel M, Cichon S, Djurovic S, Andreassen OA, Cantor RM, Ophoff R, Corvin A, Morris DW, Gill M, Pato CN, Pato MT, Macedo A, Gurling HM, McQuillin A, Pimm J, Hultman C, Lichtenstein P, Sklar P, Purcell SM, Scolnick E, St Clair D, Blackwood DH, Kendler KS; GROUP investigators; International Schizophrenia Consortium. GWA study data mining and independent replication identify cardiomyopathy-associated 5 (CMYA5) as a risk gene for schizophrenia. Mol Psychiatry. 2011 Nov;16(11):1117-29. doi: 10.1038/mp.2010.96. Epub 2010 Sep 14. PMID 20838396
- [Background] Ashbrook DG, Williams RW, Lu L, Hager R. A cross-species genetic analysis identifies candidate genes for mouse anxiety and human bipolar disorder. Front Behav Neurosci. 2015 Jul 1;9:171. doi: 10.3389/fnbeh.2015.00171. eCollection 2015. PMID 26190982
- [Background] McCalmon SA, Desjardins DM, Ahmad S, Davidoff KS, Snyder CM, Sato K, Ohashi K, Kielbasa OM, Mathew M, Ewen EP, Walsh K, Gavras H, Naya FJ. Modulation of angiotensin II-mediated cardiac remodeling by the MEF2A target gene Xirp2. Circ Res. 2010 Mar 19;106(5):952-60. doi: 10.1161/CIRCRESAHA.109.209007. Epub 2010 Jan 21. PMID 20093629
- [Background] Pison L, De Vusser P, Mullens W. Apical ballooning in relatives. Heart. 2004 Dec;90(12):e67. doi: 10.1136/hrt.2004.046813. PMID 15547001
- [Background] Kumar G, Holmes DR Jr, Prasad A. "Familial" apical ballooning syndrome (Takotsubo cardiomyopathy). Int J Cardiol. 2010 Oct 29;144(3):444-5. doi: 10.1016/j.ijcard.2009.03.078. Epub 2009 Apr 17. PMID 19375184
- [Background] Sharkey SW, Lips DL, Pink VR, Maron BJ. Daughter-mother tako-tsubo cardiomyopathy. Am J Cardiol. 2013 Jul 1;112(1):137-8. doi: 10.1016/j.amjcard.2013.02.063. Epub 2013 Apr 2. PMID 23561588
- [Background] Caretta G, Robba D, Vizzardi E, Bonadei I, Raddino R, Metra M. Tako-tsubo cardiomyopathy in two sisters: a chance finding or familial predisposition? Clin Res Cardiol. 2015 Jul;104(7):614-6. doi: 10.1007/s00392-015-0837-0. Epub 2015 Mar 6. No abstract available. PMID 25743177
- [Derived] Khan H, Rudd A, Gamble DT, Mezincescu AM, Cheyne L, Horgan G, Dhaun N, Newby DE, Dawson DK. Renin-Angiotensin and Endothelin Systems in Patients Post-Takotsubo Cardiomyopathy. J Am Heart Assoc. 2022 Jul 19;11(14):e025989. doi: 10.1161/JAHA.122.025989. Epub 2022 Jul 13. PMID 35861811
- [Derived] Scally C, Abbas H, Ahearn T, Srinivasan J, Mezincescu A, Rudd A, Spath N, Yucel-Finn A, Yuecel R, Oldroyd K, Dospinescu C, Horgan G, Broadhurst P, Henning A, Newby DE, Semple S, Wilson HM, Dawson DK. Myocardial and Systemic Inflammation in Acute Stress-Induced (Takotsubo) Cardiomyopathy. Circulation. 2019 Mar 26;139(13):1581-1592. doi: 10.1161/CIRCULATIONAHA.118.037975. PMID 30586731